CLINICAL TRIAL: NCT03760679
Title: Comparison of Laryngeal Mask Supreme and I-Gel in Edentulate Geriatric Patients
Brief Title: Laryngeal Mask Supreme and I-Gel in Edentulate Geriatric Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Sule Ozbilgin, Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 341-SBKAEK
Record Dates: First submitted 2018-08-30; First posted 2018-11-30 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Airway Morbidity
Keywords: laryngeal mask; geriatric; patient

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laryngeal mask Supreme (Active Comparator): Device: Laryngeal mask Supreme
  Interventions: Device: Laryngeal mask Supreme evaluation
- i-gel (Experimental): Device: i-gel
  Interventions: Device: i-gel evaluation

INTERVENTIONS:
Device: Laryngeal mask Supreme evaluation — Device: Laryngeal mask Supreme evaluation
  Other Names: Device: Laryngeal mask Supreme evaluation
  Arms: Laryngeal mask Supreme
Device: i-gel evaluation — Device: i-gel evaluation
  Other Names: Device: i-gel evaluation
  Arms: i-gel

SUMMARY:
The primary aim of this study is to evaluate ease and duration of placing Laryngeal Mask Supreme (LM) and applying I-gel in geriatric patients without teeth. The secondary aim is to compare their effects on ventilation parameters.

DETAILED DESCRIPTION:
Prospective, randomized and double-blind study, aged from 18 to 65 years undergoing elective laparoscopic gynecological surgery.

The patients are randomly assigned to 2 groups:

* Group 1: i-gel
* Group 2: laryngeal mask airway - Supreme

Procedure:

The investigation protocol contains the following sections:

1. Induction of anaesthesia: Preoxygenation will be provided at 6 Liter/min oxygen for three minutes by using a facial mask. After anesthesia induction with fentanyl 1-2 μg/kg and propofol 1-2 mg/kg (12), mask ventilation will be applied with 100% oxygen.
2. Bispectral index values will be held between 40-60.Bispectral index values will be within this interval by increasing or decreasing propofol infusion by 1 mg/kg after additional bolus dose of propofol (1 mg/kg).
3. Insertion of the airway device. The size of the airway device used is based on the manufacturers' recommendations. All devices are deflated a lubricated prior to use. Once inserted, the cuff is be inflated with a manometer up to 60 cm H20 Data recorded: size of airway device, time an number of attempts.
4. Maintenance of anesthesia will be achieved with sevoflurane 1,5-2,5% in a mixture of 50% O2/ 50% nitrogen protoxide. Sevoflurane concentrations will be adjusted to keep bispectral index values at 40-60.
5. Measurement of airway seal pressure (oropharyngeal leak pressure (OLP): at baseline, and two minutes after the airway tool is placed, every 15 minutes until the operation ends and before the airway tool is removed.
6. Ventilatory mechanics and parameters and hemodynamic parameters are measured at baseline, and two minutes after the airway tool is placed, every 15 minutes until the operation ends and before the airway tool is removed.
7. Perioperative complications: Cough, vomiting, laryngeal spasm, laryngeal Stridor
8. Removal of the airway device: Presence of blood - 3 level grading (1:no blood; 2: trace amounts of blood; 3: clear amounts of blood). Complications: sore throat (visual analogue scale :10-point scale), dysphonia (yes/no), dysphagia (yes/no).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Classification I-III patients
* patients aged 65 years and older

Exclusion Criteria:

* having teeth or fixed prosthesis
* having a pathology of the neck or the upper respiratory tract
* having a risk of regurgitation of gastric content/ aspiration (prior upper gastrointestinal system surgery, hiatus hernia, gastrointestinal reflux, history of peptic ulcer and full stomach)
* history or possibility of difficult airway (history of impossible intubation, mallampati score of 3-4, sternomental distance of shorter than 12 cm, thyromental distance of shorter than 6cm, head extension of lower than 90 degrees and mouth opening of lower than 1.5 cm)
* lower pulmonary compliance or higher airway resistance (morbid obesity -BMI>35kg/m2- and pulmonary disease) Each patient will be examined preoperatively and American Society of Anesthesiologists Classification scores and mallampati scores will be recorded. Standard monitoring (ECG, pulse oximetry and noninvasive blood pressure measurement) and bispectral index monitoring will be performed in each patient before induction of anesthesia in the surgical room.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Airway Seal Pressure Values | intraoperative
insertion time | intraoperative
  placement of airway device (second)

SECONDARY OUTCOMES:
sore throat | postoperative 1th hour and 24th hour
  postoperative pharyngolaryngeal morbidity- (Visual Analog Pain Scale is a unidimensional measure of pain intensity ), ("no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale])
dysphagia | postoperative 1th hour and 24th hour
  postoperative pharyngolaryngeal morbidity- dysphagia (yes/no)
dysphonia | postoperative 1th hour and 24th hour
  postoperative pharyngolaryngeal morbidity- dysphonia (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Büyükçoban, Principal Investigator — Dokuz Eylül University, School of Medicine, Department of Anesthesiology and Intensive Care
Locations (1):
- Şule Özbilgin, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided